CLINICAL TRIAL: NCT06451926
Title: The Effect of Educational Escape Room Instruction on Nursing Students' Intravenous Drug Dose Calculation and Fluid Therapy Application Skills
Brief Title: Educational Escape Room Game and Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şırnak Üniversitesi (Other)
Responsible Party: Principal Investigator, Hursit Fidan, Lecturer, Şırnak Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Şırnak University
Record Dates: First submitted 2024-05-13; First posted 2024-06-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Gamification
Keywords: Escape Room,; Nursing Students,; Drug Dosage Calculation,; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: experimental group
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): escape room game (play group):The experimental group will play the educational escape room game. The experimental group will play the game once in total.
  Interventions: Other: Escape room game
- Control (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Other: Escape room game — Educational escape rooms are live action games where teams use content knowledge to complete tasks and puzzles to reach a final goal, such as escaping from a room or completing a final puzzle
  Arms: Experimental

SUMMARY:
This study will be conducted to determine the effect of educational escape room teaching on nursing students' skills in calculating intravenous drug dosage and applying fluid therapy. The research was planned in a pretest-posttest and retest randomized controlled experimental design with a control group.

This study will be conducted in the Spring Term of the 2023-2024 Academic Year at Kafkas University, Faculty of Health Sciences, Department of Nursing. 1st year and 4th year nursing students will be included in the sample of the research.

Power analysis was performed to determine the number of people to be included in the study. The power of the test was calculated with the G*Power 3.1 program. Students will be divided into two groups, control and experimental, by randomization method. A total of 120 students were planned to be included in the study: 30 experimental and 30 control students for the first grade, and 30 experimental and 30 control students for the fourth grade.

In order to conduct the research, written permissions were obtained from the ethics committee and the institution where the study would be conducted.

The data of the research will be collected with the "Introductory Information Form-IIF", "Intravenous Drug Dosage Calculation and Fluid Therapy Application Knowledge Test-IVKT" (min:0-max:100), "Intravenous Drug Dosage Calculation and Fluid Therapy Application Skill Checklists-IVSC" (min:0-max:242) and "Game Evaluation Form-GEF" (min:26-max:130). Increasing the score obtained from data collection tools means that knowledge and skills increase.Data collection tools were presented to expert opinion for content validity. Content validity indexes were calculated and it was determined that the instruments were usable. The entire sample group will be given training on intravenous drug dose calculation and fluid therapy application. During the training, the subject will be supported by question-answer technique. Then, initial knowledge (pre-test) and initial skill (pre-test) will be measured with an objective structured clinical exam and scores will be calculated. According to the pre-test knowledge and skill scores, students from both grade levels will be assigned to experimental and control groups. The experimental group will play the escape room game in teams of five people according to the prepared educational escape room game plan. During this process, the control group will be given the right to work independently in the laboratory. The experimental group will play the educational escape room game once, and then the final knowledge (post-test) and final skills (objective structured clinical exam) of the experimental and control groups will be measured. Each student in the experimental group will be asked to fill out the game evaluation form.

In evaluating the data, parametric or non-parametric tests will be used to determine whether the research data show a normal distribution or not. Correlation will be made to determine the relationship between pretest and posttest knowledge tests and objective structured clinical exam scores. Regression analysis will also be performed if necessary, based on the analysis results of the research data.

DETAILED DESCRIPTION:
In the sample group, the first knowledge (pre-test) scores will be measured after the training of intravenous drug dose calculation and fluid therapy application training and question-answer. First skill (pre-test) scores will be measured with objective structured clinical exam.

Students' skills will be evaluated by independent observers other than researchers, using checklists, through the objective structured clinical exam exam. Then, students will be assigned to experimental and control groups by randomization according to their initial knowledge and skill scores.

The "educational escape room" game prepared by researchers in the faculty's nursing skills laboratory will be played to the experimental groups once on different days. Then, the "Game Evaluation Form-GEF" will be applied to the experimental groups. In this process, the control group will be given the right to work independently in another skill laboratory of the faculty to perform the relevant skills.

After the educational escape room game, the final knowledge of both the experimental and control groups will be measured again (post-test). All students' skills will then be measured by independent observers through the objective structured clinical exam (post-test). Two weeks after the post-test, the knowledge and skill (objective structured clinical exam) scores of the students will be measured.

Experimental groups will play the educational escape room game once. The game will take place in a total of three rooms. In each room, there are a total of five patient scenarios that will require students to perform different skills individually and a total of five game activities (puzzles, jigsaws, etc.) to be performed by the team. They will enter the rooms in order, each student will perform the skill in the scenario for which they are responsible, and then they will perform the game activity they need to perform as a team. After each game event they will receive a number code needed to escape the clinic. They will finish the game by opening the five number codes they obtained in this way and the locked box with the number code.

Educational escape room game is a type of game in which groups of four to ten people work together and learn to complete some game activities in order to escape from a locked room in a limited time period. This game, in which students use communication, collaboration and critical thinking skills while learning, has recently begun to be used frequently in the field of education and training.

ELIGIBILITY:
Inclusion criteria:

* Volunteering to participate in the research,
* Being a first year nursing student,
* Being a fourth year nursing student
* First-year nursing students must be enrolled in the Fundamentals of Nursing II course,
* Fourth year nursing students must have taken the Fundamentals of Nursing II course,

Exclusion Criteria:

* Not participating in the training program,
* Not wanting to continue research,
* Incomplete filling of data collection tools,
* Incorrect filling of data collection tools,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Measuring the knowledge level of the sample group | Pre-test data will be collected in the first week of implementation (before randomization).
  The knowledge levels of all students who will participate in the study will be measured with the 'Intravenous Drug Dose Calculation and Fluid Therapy Application Knowledge Test'.
Measuring the skill levels of the sample group | Pre-test data will be collected in the first week of implementation(before randomization).
  The skill levels of all students who will participate in the study will be measured with 'Intravenous Drug Dose Calculation and Fluid Therapy Application Skill Checklists.

SECONDARY OUTCOMES:
Measurement of knowledge levels of experimental and control groups | Post-test data will be collected after the educational escape game in the second week of the application (post escape room game).
  The experimental group will play the educational escape room game once and then the final knowledge (post-test) of the experimental and control groups will be measured with the 'Intravenous Drug Dose Calculation and Fluid Therapy Application Knowledge Test'.
Measuring the skills of the experimental and control groups | Post-test data will be collected after the educational escape game in the second week of the application (post escape room game).
  The experimental group will play the educational escape room game once and then the final knowledge (post-test) of the experimental and control groups will be measured with the 'Intravenous Drug Dose Calculation and Fluid Therapy Application Skill Checklists'.

OTHER OUTCOMES:
Retest of skills and knowledge levels of experimental and control groups | The test will be repeated two weeks after the post-test.
  The retest knowledge and skills of the experimental and control groups will be measured with 'Intravenous Drug Dose Calculation and Fluid Therapy Application Skill Checklists' and 'Intravenous Drug Dose Calculation and Fluid Therapy Application Knowledge Test' two weeks after the educational escape room game was played (retest).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafkas University Faculty of Health Sciences, Kars, Centre/Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No